CLINICAL TRIAL: NCT05605613
Title: PD-1 Antibody in Addition to Bronchial Arterial Chemoembolization in Patients With Non-Small-Cell Lung Cancer: A Randomised Controlled Trial
Brief Title: PD-1 Antibody in Addition to BACE in Patients With NSCLC: A Randomised Controlled Trial
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuhua Duan (Other)
Responsible Party: Sponsor-Investigator, Xuhua Duan, Associate Professor, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20221030
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: NSCLC
Keywords: BACE; PD-1 Antibody
MeSH Terms: interventions — spartalizumab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-1 Antibody in Addition to Bronchial Arterial Chemoembolization (Experimental): Treated with BACE and PD-1 antibody as induction therapy during which BACE was performed on the first day and PD-1 antibody was given 3-5 days later, then PD-1 antibody was administered at 200mg Q3W as maintenance therapy.
  Interventions: Drug: PD-1 Antibody; Device: BACE
- Bronchial Arterial Chemoembolization (Active Comparator): Bronchial artery chemoembolization (BACE) is a technique of drug delivery and embolization performed via injecting anti-tumor drugs with drug carriers and implanting the embolization agents into the tumor feeding artery
  Interventions: Device: BACE

INTERVENTIONS:
Drug: PD-1 Antibody — PD-1 Antibody, an investigational humanized IgG4 monoclonal antibody with high affinity and binding specificity for PD-1
  Other Names: PD-1 Inhibitors
  Arms: PD-1 Antibody in Addition to Bronchial Arterial Chemoembolization
Device: BACE — Bronchial Arterial Chemoembolization

SUMMARY:
This is a randomized controlled trial to determine the efficacy and safety of PD-1 Antibody in addition to Bronchial Arterial Chemoembolization in stage III-Ⅳ NSCLC patients who failed, refused or ineligible to receive standard treatments.

DETAILED DESCRIPTION:
Bronchial artery chemoembolization (BACE) is a technique of drug delivery and embolization performed via injecting anti-tumor drugs with drug carriers and implanting the embolization agents into the tumor feeding artery, promoting the clinical outcomes of patients and providing a palliative treatment option for patients with NSCLC. while the short-term effect of BACE is good, it is easy to relapse and metastasize.

The rapid development of immunotherapy checkpoint inhibitors represented by PD-1/L1 monoclonal antibody has changed the treatment pattern of NSCLC. The publication of early research data repeatedly verified the long-term survival benefit characteristics of PD-1/L1 in NSCLC.

Based on this research and clinical practice, we designed this trial to determine the efficacy and safety of PD-1 antibody in addition to Bronchial Arterial Chemoembolization in stage III-Ⅳ NSCLC patients who failed, refused or ineligible to receive standard treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age between 18 and 75
2. Signed Informed Consent Form.
3. Confirmed TNM stage is III-Ⅳ of NSCLC ，and failed, refused or assessed ineligible to receive conventional treatments (surgery, chemoradiotherapy, chemotherapy )； Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
4. Adequate hematologic and end-organ function.
5. Expected life span > 3 months.
6. Be able to provide fresh or archival tumor tissues for PD-L1 expression in tumor cells

Exclusion Criteria:

1. Prior treatment targeting PD-1, PD-L1 or CTLA-4.
2. Prior therapies of interventional therapy (I seed implantation, Ablation, BACE).
3. Harboring EGFR sensitizing mutation or ALK gene translocation
4. History of interstitial lung disease, non-infectious pneumonitis or participants with significantly impaired pulmonary function, or who require supplemental oxygen at baseline.
5. With uncontrollable pleural effusion, pericardial effusion, or clinically significant ascites requiring interventional treatment.
6. Symptomatic central nervous system metastasis
7. Known HIV infection, participants with untreated chronic hepatitis B, active vaccination treatment.
8. Prior allogeneic stem cell transplantation or organ transplantation
9. Active autoimmune diseases or history of autoimmune diseases that may relapse.
10. With conditions requiring systemic treatment with either corticosteroids (>10 mg daily prednisone or equivalent) or other immunosuppressive medications
11. Known to be hypersensitive to contrast agent;
12. Pregnant or breastfeeding women;
13. Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-10-29 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Time from the first BACE treatment to either radiological progression or death or up to 12 months]
  Time from the first BACE treatment to either radiological progression or death

SECONDARY OUTCOMES:
Objective response rate (ORR) | Time Frame: 2, 4, 6 months after the first BACE treatment, up to death or 12 months
  Proportion of patients with reduction in stable in tumor burden of a predefined amount
Disease control rate (DCR) | 2, 4, 6 months after the first BACE treatment, up to death or 12 months
  Proportion of patients with reduction or keeping in stable in tumor burden of a predefined amount
Overall survival (OS) | 1 years
  ime from the first BACE treatment to death from any cause or the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Xuhua Duan, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (8):
- China (8):
  - People's Hospital of Kaiyang County, Guiyang, Guizhou
  - North China University of Science and Technology Affiliated Hospital, Tangshan, Hebei
  - The Second Affiliated Hospital of Xingtai Medical College, Xingtai, Hebei
  - Hebi City Jun County People's Hospital, Hebi, Henan
  - Wuyang County People's Hospital, Luohe, Henan
  - Dengzhou People's Hospital, Nanyang, Henan
  - The Fifth People's Hospital of Puyang City, Puyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan